CLINICAL TRIAL: NCT02284152
Title: Responsive Feeding Study
Acronym: RFS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: Monell Chemical Senses Center (Other)
Responsible Party: Principal Investigator, Alison Ventura, Assistant Professor, Drexel University
Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 809649
Record Dates: First submitted 2014-11-03; First posted 2014-11-05 (Estimated); Last update posted 2014-11-05 (Estimated); Status verified 2014-11

CONDITIONS: Bottle Feeding
Keywords: bottle feeding; feeding behavior; infants; mothers; responsive feeding; maternal feeding practices; maternal feeding styles
MeSH Terms: conditions — Bottle Feeding; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Typical versus Infant-Led feeding (Experimental): This is a within-subject study; all infants and mothers will be exposed to both conditions (typical feeding versus infant-led feeding conditions). Order of presentation will be counterbalanced across infant/mother dyads.
  Interventions: Behavioral: infant-led feeding

INTERVENTIONS:
Behavioral: infant-led feeding — mothers' feeding practices and infant intakes were compared between a typical feeding condition and an infant-led feeding condition, where the experimenter ensured the feeding was in response to infant hunger and fullness cues.

SUMMARY:
In the present study, we tested a novel approach to understanding infant bottle-feeding interactions: experimentally manipulating bottle-feeding conditions to better understand maternal and infant influences on overfeeding, as well as individual differences in risk for overfeeding. Specifically, we observed mother-infant dyads during a typical, "mother-led" feeding, during which mothers were given no instruction regarding how or how much to feed their infants (hereafter referred to as a "typical feeding" [TF]), as well as during an "infant-led" (IL) feeding, wherein we minimized the mothers' influence on the feeding and ensured the feed was in response to the infants' hunger and fullness cues. Using this within-subject, objective, and experimental approach, the present study aimed to: 1) directly measure the extent to which overfeeding occurs during bottle-feeding and 2) describe the characteristics of infants and mothers that overfeed during bottle-feeding.

DETAILED DESCRIPTION:
Each mother-infant dyad came to our laboratory on two different days, separated by an average of 2.1 ± 0.4 days. The two testing sessions occurred at the same time of day to control for infants' circadian rhythmicity. Mothers were instructed to bring two of their infants' typical bottles filled with their infants' typical formula to each testing session. Mothers were videotaped while feeding their infants on both days. The first day of testing was always the Typical Feeding (TF) condition because the only instruction given to the mother was: "Please feed your infant as you normally would at home." The second day of testing was always the Infant-Led (IL) condition, wherein we used a protocol developed and established in our laboratory to control for a number of factors to allow for evaluation of infants' hedonic and behavioral responses independent of the parent and experimenter. The feeding protocol during the IL condition entailed the following steps, which were facilitated by the experimenter: (1) feeding sessions began when the experimenter observed the infant displaying signs of hunger (e.g., mouthing, rooting, fussing) and the mother verified that the infant was hungry; (2) the mother was instructed not to talk to her infant and to remain as neutral as possible; (3) the mother was also instructed to feed her infant at his/her customary pace; (4) the experimenter ended the feeding when the infant displayed signs of fullness (e.g., turning head and/or body away from the bottle, biting or chewing on the nipple, spiting the nipple out) on at least three consecutive occasions. If the infant finished the bottle before signaling fullness, the experimenter gave the mother the other bottle to ensure that infant intake was not limited by formula availability. During both study days, consumption during the feeding session was assessed by weighing the bottles before and after each feeding using a top loading balance (model PM 15; Mettler, Greifensee, Switzerland).

ELIGIBILITY:
Inclusion Criteria:

* Formula-feeding
* Prior to the introduction of solid foods
* Infants 0 to 6 months of age
* Mothers 18 to 40 years of age

Exclusion Criteria:

* Exclusively breast-feeding
* Preterm
* Medical conditions that interfered with feeding

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Infant Intake | 3-hour period
  Infant intake was assessed by weighing the bottle before and after the feeding

CONTACTS AND LOCATIONS:
Overall Officials: Alison K Ventura, PhD, Principal Investigator — Cal Poly University
Locations (3):
- United States (3):
  - California Polytechnic State University, San Luis Obispo, California
  - Drexel University, Philadelphia, Pennsylvania
  - Monell Chemical Senses Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Ventura AK, Inamdar LB, Mennella JA. Consistency in infants' behavioural signalling of satiation during bottle-feeding. Pediatr Obes. 2015 Jun;10(3):180-7. doi: 10.1111/ijpo.250. Epub 2014 Jul 3. PMID 24990443